CLINICAL TRIAL: NCT04070456
Title: Addressing Social Determinants of Health to Reduce Physician Burnout
Brief Title: Clinician Burnout and Social Determinants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00059798; 1902014 (Other Grant/Funding Number: American Medical Association)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-06

CONDITIONS: Burnout, Professional
Keywords: Physician Burnout; social determinants of health; Mini-Z
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention sites-Tablet-based SDH tool (Experimental): All clinicians and primary care teams at a practice that are randomized to the intervention will receive the tablet-based SDH tool.
  Interventions: Other: Tablet-based SDH tool
- Control sites (No Intervention): Care as usual, no tablet-based SDH tool.

INTERVENTIONS:
Other: Tablet-based SDH tool — A tablet-based SDH tool, which integrates responses into the EpicCare electronic health record (EHR).
  Arms: Intervention sites-Tablet-based SDH tool

SUMMARY:
Although clinicians recognize the impact of the social determinants of health (SDH) on patient care, clinicians feel they do not have the time or knowledge to effectively address patients' unmet social needs in the clinic. This can lead to feelings of distress and helplessness. The objective of this study is to test the impact of a tablet-based platform that enhances the role of support staff to address SDH on clinician burnout.

DETAILED DESCRIPTION:
Clinician burnout has risen over the last decade, and studies have found that almost 50% of U.S. physicians show signs of burnout. Burnout is characterized by emotional exhaustion, feelings of cynicism, and patient detachment. Clinicians at the front lines of care, such as family medicine and internal medicine, are at highest risk, and burnout is associated with an increased risk of cardiovascular disease, alcoholism, and suicide. Burnout also negatively impacts patient care. The drivers of burnout are complex, and a growing body of research has focused on developing strategies to address both clinician and organizational factors. One potential contributor to clinician burnout that has received less attention is their patients' SDH.

The SDH, or the circumstances in which people are born, grow, live, and age, have a profound impact on morbidity and mortality. Increasingly, national organizations have called for healthcare systems to address SDH, such as food and housing insecurity, to improve population health. Although clinicians recognize the importance of SDH on patient care, clinicians feel they do not have the time, knowledge, or tools to effectively address SDH, which can leading to feelings of distress and helplessness in addressing patients' unmet social needs. The SDH can lead to increased patient complexity and clinician workload. Also, the seemingly insurmountable social needs faced by many patients are a major contributor to the decline in medicine residents choosing a career in primary care. Thus, the lack of a tool to assist the primary care team in addressing SDH is a critical problem that can negatively affect both patients and clinicians.

Our long-term goal is to enhance the primary care teams' ability to address the SDH by utilizing a mobile health tool that can assist the team in addressing patients' unmet social needs in clinical settings. Mobile health tools, such as tablets, have shown promise in reducing disparities in care and addressing unmet social needs in pediatric practices. However, there is little data about how addressing SDH affects physician burnout. Mobile health tools have the potential to collect patient-reported data and connect patients to appropriate support personnel without interfering with clinic workflow and enhance the primary care teams' ability to provide patients with resources. The objective of this study is to test the impact of a tablet-based platform that enhances the role of support staff to address SDH on clinician burnout.

ELIGIBILITY:
Inclusion Criteria:

* All clinicians and primary care teams at participating sites will be eligible

Exclusion Criteria:

* There are no specific exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Mini-Z Scale | Baseline
  This scales measures clinician satisfaction. Total score 10 to 45. Higher scores denotes better outcome.
Mini-Z Scale | 6 month post baseline
  This scales measures clinician satisfaction. Total score 10 to 45. Higher scores denotes better outcome.
Mini-Z Scale | 12 month post baseline
  This scales measures clinician satisfaction. Total score 10 to 45. Higher scores denotes better outcome.

SECONDARY OUTCOMES:
The number of clinicians who report a joyful workplace | Baseline
The number of clinicians who report a joyful workplace | 6 months post baseline
The number of clinicians who report a joyful workplace | 12 months post baseline
The number of clinicians who report a supportive practice | Baseline
The number of clinicians who report a supportive practice | 6 months post baseline
The number of clinicians who report a supportive practice | 12 months post baseline
The number of clinicians who report a good work pace | Baseline
The number of clinicians who report a good work pace | 6 months post baseline
The number of clinicians who report a good work pace | 12 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Palakshappa, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Wake Forest Downtown Health Plaza (DHP), Winston-Salem, North Carolina
  - Family Medicine-Piedmont Plaza, Winston-Salem, North Carolina
  - Internal Medicine-Janeway Tower, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deindentification
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication, no end date
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Background] Shanafelt TD, Boone S, Tan L, Dyrbye LN, Sotile W, Satele D, West CP, Sloan J, Oreskovich MR. Burnout and satisfaction with work-life balance among US physicians relative to the general US population. Arch Intern Med. 2012 Oct 8;172(18):1377-85. doi: 10.1001/archinternmed.2012.3199. PMID 22911330
- [Background] Shanafelt TD, Hasan O, Dyrbye LN, Sinsky C, Satele D, Sloan J, West CP. Changes in Burnout and Satisfaction With Work-Life Balance in Physicians and the General US Working Population Between 2011 and 2014. Mayo Clin Proc. 2015 Dec;90(12):1600-13. doi: 10.1016/j.mayocp.2015.08.023. PMID 26653297
- [Background] Shanafelt TD, Noseworthy JH. Executive Leadership and Physician Well-being: Nine Organizational Strategies to Promote Engagement and Reduce Burnout. Mayo Clin Proc. 2017 Jan;92(1):129-146. doi: 10.1016/j.mayocp.2016.10.004. Epub 2016 Nov 18. PMID 27871627
- [Background] C M, S J, M L. Maslach Burnout Inventory Manual. Consulting Psychologist Press. 1996;3rd edition.
- [Background] Shanafelt TD, Balch CM, Dyrbye L, Bechamps G, Russell T, Satele D, Rummans T, Swartz K, Novotny PJ, Sloan J, Oreskovich MR. Special report: suicidal ideation among American surgeons. Arch Surg. 2011 Jan;146(1):54-62. doi: 10.1001/archsurg.2010.292. PMID 21242446
- [Background] Shanafelt TD, Balch CM, Bechamps G, Russell T, Dyrbye L, Satele D, Collicott P, Novotny PJ, Sloan J, Freischlag J. Burnout and medical errors among American surgeons. Ann Surg. 2010 Jun;251(6):995-1000. doi: 10.1097/SLA.0b013e3181bfdab3. PMID 19934755
- [Background] Shanafelt TD, Gradishar WJ, Kosty M, Satele D, Chew H, Horn L, Clark B, Hanley AE, Chu Q, Pippen J, Sloan J, Raymond M. Burnout and career satisfaction among US oncologists. J Clin Oncol. 2014 Mar 1;32(7):678-86. doi: 10.1200/JCO.2013.51.8480. Epub 2014 Jan 27. PMID 24470006
- [Background] Panagioti M, Geraghty K, Johnson J, Zhou A, Panagopoulou E, Chew-Graham C, Peters D, Hodkinson A, Riley R, Esmail A. Association Between Physician Burnout and Patient Safety, Professionalism, and Patient Satisfaction: A Systematic Review and Meta-analysis. JAMA Intern Med. 2018 Oct 1;178(10):1317-1331. doi: 10.1001/jamainternmed.2018.3713. PMID 30193239 (Retraction: PMID 32421149 JAMA Intern Med. 2020 Jul 1;180(7):931)
- [Background] Shanafelt TD, Dyrbye LN, West CP, Sinsky CA. Potential Impact of Burnout on the US Physician Workforce. Mayo Clin Proc. 2016 Nov;91(11):1667-1668. doi: 10.1016/j.mayocp.2016.08.016. No abstract available. PMID 27814840
- [Background] Shanafelt TD, Mungo M, Schmitgen J, Storz KA, Reeves D, Hayes SN, Sloan JA, Swensen SJ, Buskirk SJ. Longitudinal Study Evaluating the Association Between Physician Burnout and Changes in Professional Work Effort. Mayo Clin Proc. 2016 Apr;91(4):422-31. doi: 10.1016/j.mayocp.2016.02.001. PMID 27046522
- [Background] Dyrbye LN, Trockel M, Frank E, Olson K, Linzer M, Lemaire J, Swensen S, Shanafelt T, Sinsky CA. Development of a Research Agenda to Identify Evidence-Based Strategies to Improve Physician Wellness and Reduce Burnout. Ann Intern Med. 2017 May 16;166(10):743-744. doi: 10.7326/M16-2956. Epub 2017 Apr 18. No abstract available. PMID 28418518
- [Background] Eisenstein L. To Fight Burnout, Organize. N Engl J Med. 2018 Aug 9;379(6):509-511. doi: 10.1056/NEJMp1803771. Epub 2018 Jun 20. No abstract available. PMID 29924700
- [Background] Byhoff E, Freund KM, Garg A. Accelerating the Implementation of Social Determinants of Health Interventions in Internal Medicine. J Gen Intern Med. 2018 Feb;33(2):223-225. doi: 10.1007/s11606-017-4230-8. Epub 2017 Nov 29. No abstract available. PMID 29188543
- [Background] Long T, Chaiyachati K, Bosu O, Sircar S, Richards B, Garg M, McGarry K, Solomon S, Berman R, Curry L, Moriarty J, Huot S. Why Aren't More Primary Care Residents Going into Primary Care? A Qualitative Study. J Gen Intern Med. 2016 Dec;31(12):1452-1459. doi: 10.1007/s11606-016-3825-9. Epub 2016 Aug 3. PMID 27488970
- [Background] Gottlieb LM, Francis DE, Beck AF. Uses and Misuses of Patient- and Neighborhood-level Social Determinants of Health Data. Perm J. 2018;22:18-078. doi: 10.7812/TPP/18-078. PMID 30227912
- [Background] Chetty R, Stepner M, Abraham S, Lin S, Scuderi B, Turner N, Bergeron A, Cutler D. The Association Between Income and Life Expectancy in the United States, 2001-2014. JAMA. 2016 Apr 26;315(16):1750-66. doi: 10.1001/jama.2016.4226. PMID 27063997
- [Background] Gottlieb LM, Wing H, Adler NE. A Systematic Review of Interventions on Patients' Social and Economic Needs. Am J Prev Med. 2017 Nov;53(5):719-729. doi: 10.1016/j.amepre.2017.05.011. Epub 2017 Jul 5. PMID 28688725
- [Background] Marmot M, Shipley M, Brunner E, Hemingway H. Relative contribution of early life and adult socioeconomic factors to adult morbidity in the Whitehall II study. J Epidemiol Community Health. 2001 May;55(5):301-7. doi: 10.1136/jech.55.5.301. PMID 11297647
- [Background] Marmot MG, Bosma H, Hemingway H, Brunner E, Stansfeld S. Contribution of job control and other risk factors to social variations in coronary heart disease incidence. Lancet. 1997 Jul 26;350(9073):235-9. doi: 10.1016/s0140-6736(97)04244-x. PMID 9242799
- [Background] Alley DE, Asomugha CN, Conway PH, Sanghavi DM. Accountable Health Communities--Addressing Social Needs through Medicare and Medicaid. N Engl J Med. 2016 Jan 7;374(1):8-11. doi: 10.1056/NEJMp1512532. Epub 2016 Jan 5. No abstract available. PMID 26731305
- [Background] Garg A, Boynton-Jarrett R, Dworkin PH. Avoiding the Unintended Consequences of Screening for Social Determinants of Health. JAMA. 2016 Aug 23-30;316(8):813-4. doi: 10.1001/jama.2016.9282. No abstract available. PMID 27367226
- [Background] Garg A, Jack B, Zuckerman B. Addressing the social determinants of health within the patient-centered medical home: lessons from pediatrics. JAMA. 2013 May 15;309(19):2001-2. doi: 10.1001/jama.2013.1471. No abstract available. PMID 23619825
- [Background] Nuruzzaman N, Broadwin M, Kourouma K, Olson DP. Making the social determinants of health a routine part of medical care. J Health Care Poor Underserved. 2015 May;26(2):321-7. doi: 10.1353/hpu.2015.0036. No abstract available. PMID 25913331
- [Background] Services USDoHaH. HealthyPeople 2020. 2017; https://http://www.healthypeople.gov/2020/topics-objectives/topic/nutrition-and-weight-status. Accessed Sept 30, 2017.
- [Background] DeVoe JE, Bazemore AW, Cottrell EK, Likumahuwa-Ackman S, Grandmont J, Spach N, Gold R. Perspectives in Primary Care: A Conceptual Framework and Path for Integrating Social Determinants of Health Into Primary Care Practice. Ann Fam Med. 2016 Mar;14(2):104-8. doi: 10.1370/afm.1903. No abstract available. PMID 26951584
- [Background] Gottlieb L, Hessler D, Long D, Amaya A, Adler N. A randomized trial on screening for social determinants of health: the iScreen study. Pediatrics. 2014 Dec;134(6):e1611-8. doi: 10.1542/peds.2014-1439. Epub 2014 Nov 3. PMID 25367545
- [Background] Hassan A, Scherer EA, Pikcilingis A, Krull E, McNickles L, Marmon G, Woods ER, Fleegler EW. Improving Social Determinants of Health: Effectiveness of a Web-Based Intervention. Am J Prev Med. 2015 Dec;49(6):822-31. doi: 10.1016/j.amepre.2015.04.023. Epub 2015 Jul 26. PMID 26215831
- [Background] Wu S, Ell K, Jin H, Vidyanti I, Chou CP, Lee PJ, Gross-Schulman S, Sklaroff LM, Belson D, Nezu AM, Hay J, Wang CJ, Scheib G, Di Capua P, Hawkins C, Liu P, Ramirez M, Wu BW, Richman M, Myers C, Agustines D, Dasher R, Kopelowicz A, Allevato J, Roybal M, Ipp E, Haider U, Graham S, Mahabadi V, Guterman J. Comparative Effectiveness of a Technology-Facilitated Depression Care Management Model in Safety-Net Primary Care Patients With Type 2 Diabetes: 6-Month Outcomes of a Large Clinical Trial. J Med Internet Res. 2018 Apr 23;20(4):e147. doi: 10.2196/jmir.7692. PMID 29685872
- [Background] Matthew-Maich N, Harris L, Ploeg J, Markle-Reid M, Valaitis R, Ibrahim S, Gafni A, Isaacs S. Designing, Implementing, and Evaluating Mobile Health Technologies for Managing Chronic Conditions in Older Adults: A Scoping Review. JMIR Mhealth Uhealth. 2016 Jun 9;4(2):e29. doi: 10.2196/mhealth.5127. PMID 27282195
- [Background] Clark DO, Srinivas P, Bodke K, Keith N, Hood S, Tu W. Addressing people and place microenvironments in weight loss disparities (APP-Me): Design of a randomized controlled trial testing timely messages for weight loss behavior in low income Black and White Women. Contemp Clin Trials. 2018 Apr;67:74-80. doi: 10.1016/j.cct.2018.01.006. Epub 2018 Jan 31. PMID 29357313
- [Background] Graham GN, Ostrowski M, Sabina AB. Population health-based approaches to utilizing digital technology: a strategy for equity. J Public Health Policy. 2016 Nov;37(Suppl 2):154-166. doi: 10.1057/s41271-016-0012-5. PMID 27899799
- [Background] Kaufman A. Theory vs Practice: Should Primary Care Practice Take on Social Determinants of Health Now? Yes. Ann Fam Med. 2016 Mar;14(2):100-1. doi: 10.1370/afm.1915. No abstract available. PMID 26951582
- [Background] Lyles CR, Altschuler A, Chawla N, Kowalski C, McQuillan D, Bayliss E, Heisler M, Grant RW. User-Centered Design of a Tablet Waiting Room Tool for Complex Patients to Prioritize Discussion Topics for Primary Care Visits. JMIR Mhealth Uhealth. 2016 Sep 14;4(3):e108. doi: 10.2196/mhealth.6187. PMID 27627965
- [Background] Patel V, Hale TM, Palakodeti S, Kvedar JC, Jethwani K. Prescription Tablets in the Digital Age: A Cross-Sectional Study Exploring Patient and Physician Attitudes Toward the Use of Tablets for Clinic-Based Personalized Health Care Information Exchange. JMIR Res Protoc. 2015 Oct 19;4(4):e116. doi: 10.2196/resprot.3806. PMID 26481906
- [Background] Linzer M, Poplau S, Babbott S, Collins T, Guzman-Corrales L, Menk J, Murphy ML, Ovington K. Worklife and Wellness in Academic General Internal Medicine: Results from a National Survey. J Gen Intern Med. 2016 Sep;31(9):1004-10. doi: 10.1007/s11606-016-3720-4. Epub 2016 May 2. PMID 27138425
- [Background] Miller DP Jr, Denizard-Thompson N, Weaver KE, Case LD, Troyer JL, Spangler JG, Lawler D, Pignone MP. Effect of a Digital Health Intervention on Receipt of Colorectal Cancer Screening in Vulnerable Patients: A Randomized Controlled Trial. Ann Intern Med. 2018 Apr 17;168(8):550-557. doi: 10.7326/M17-2315. Epub 2018 Mar 13. PMID 29532054
- [Background] Miller DP Jr, Weaver KE, Case LD, Babcock D, Lawler D, Denizard-Thompson N, Pignone MP, Spangler JG. Usability of a Novel Mobile Health iPad App by Vulnerable Populations. JMIR Mhealth Uhealth. 2017 Apr 11;5(4):e43. doi: 10.2196/mhealth.7268. PMID 28400354
- [Background] Denizard-Thompson NR, Singh S, Stevens SR, Miller DP, Wofford JL. iPod technology for teaching patients about anticoagulation: a pilot study of mobile computer-assisted patient education. Prim Health Care Res Dev. 2012 Jan;13(1):42-7. doi: 10.1017/S146342361100034X. Epub 2011 Aug 22. PMID 21854695

DOCUMENTS (1):
  • Informed Consent Form (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT04070456/ICF_000.pdf